CLINICAL TRIAL: NCT04637347
Title: Comparaison Between Ultrasound-guided Supraclavicular and Infraclavicular Approaches for Subclavian Venous Catheterization in Intensive Care Unit
Brief Title: SC vs IC Approach for US-guided SC Vein Catheterization
Acronym: USIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Trabelsi Becem, associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CIS UTSCVC
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Central Venous Catheter

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP-ISV (Other): In plane infraclavicular subclavian vein catheterization
  Interventions: Device: Catheterization approach
- IP-SSV (Other): In plane supraclavicular subclavian vein catetherization
  Interventions: Device: Catheterization approach

INTERVENTIONS:
Device: Catheterization approach — In plane infraclavicular subclavian vein VS in plane supraclavicular subclavian vein catetherization

SUMMARY:
Patients were randomly divided into two groups: ultrasound-guided (US-guided) in-plane infraclavicular subclavian vein (IP-ISV) and in-plane supraclavicular subclavian vein (IP-SSV) catheterization.

For IP-ISV cannulation, a linear transducer is placed in the infraclavicular fossa. After obtaining a long-axis view of the axillary vein and distal subclavian vein ,the needle is inserted in the midpoint of the small footprint transducer. Then,the needle is advanced under real-time US guidance until visualizing the tip of the needle inside the vein while noticing the lung pleura underneath the vessels.

For IP-SSV cannulation, a short-axis view of the IJV is obtained first. The probe is slid caudally following the IJV until getting the best long-axis view of the SCV. Using an in-plane approach, the needle is inserted at the base of the transducer at a 30° angle and advanced under the long axis under real-time US guidance targeting the SCV.

DETAILED DESCRIPTION:
Patients were randomly divided into two groups: ultrasound-guided (US-guided) in-plane infraclavicular subclavian vein (IP-ISV) and in-plane supraclavicular subclavian vein (IP-SSV) catheterization.

For IP -ISV, the Linear transducer is placed perpendicularly and inferior to clavicle. Transverse (short axis) view of subclavian vein (SCV), subclavian artery (SCA) and pleura is first obtained. With SCV centrally positioned, the transducer is rotated 90° clockwise until longitudinal view of subclavian vein is obtained. Pulse-wave Doppler view of the SCV confirms non-pulsatile flow and identifies the vessel. The needle is than inserted in the midpoint of the small footprint transducer using the in-plane approach. The needle is advanced slowly, under real-time US guidance targeting the SCV, taking note of the lung pleura underneath the vessels.

For IP-SSV cannulation, a short-axis view of the IJV is first obtained . The probe is slid caudally following the IJV until the junction of the subclavian vein (SCV) and IJV is reached in the supraclavicular fossa. The probe is then turned slightly and tilted anteriorly to get the best long-axis view of the SCV and the brachiocephalic vein .

Using an in-plane approach, the needle attached to a syringe is inserted at the base of the transducer at a 30° angle and advanced strictly under the long axis of the US probe from lateral to medial. The needle point is then guided.

In both groups, catheterization was done through Seldinger technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit requiring a central venous catheter (CVC)

Exclusion Criteria:

* Major blood coagulation disorders,
* Any thrombotic formations within the vein,
* Congenital or acquired deformity of neck or clavicle
* Cannulation site infection, hematoma and surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The overall access time | During the venous cannulation procedure
  Time from the ultrasound scanning to the ultrasound confirmation of the correct position of the guidewire into vein.
The guidewire time | During the venous cannulation procedure
  Time from the first skin puncture to the ultrasound confirmation of the correct placement of the guidewire into the vein
The venous access time | During the venous cannulation procedure
  he time between the first skin puncture and free aspiration of venous blood in the syringe

CONTACTS AND LOCATIONS:
Overall Officials: BEN ALI MECHAAL, PROFESSOR, Study Chair — University Tunis El Manar
Locations (1):
- Mrezga Nabeul Tunisie, Nabeul, Tunisia